CLINICAL TRIAL: NCT03545542
Title: Investigating the Microbiome and Volatile Organic Compound Profile of Children With Neuroblastoma - a Pilot Study
Brief Title: Investigating the Microbiome and Volatile Organic Compound Profile of Children With Neuroblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0001
Record Dates: First submitted 2018-05-07; First posted 2018-06-04 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Microbial Colonization; Neuroblastoma; Children, Only
Keywords: Microbiome; Volatile organic compounds; Neuroblastoma
MeSH Terms: conditions — Communicable Diseases; Neuroblastoma

STUDY DESIGN:
Intervention Model Description: Neuroblastoma group: Children with neuroblastoma enrolled after verification of diagnosis. Sampling before initiation of chemotherapy and under chemotherapy.
  Control group: healthy children without gastro-intestinal or pulmonary disease recruited from paediatric surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroblastoma group (Experimental): 10 children with neuroblastoma. Inclusion after verification of diagnosis and informed consent.
  Sampling of fecal microbiome (Initial microbiome, microbiome under chemotherapy, final microbiome), fecal volatile organic compounds (initial fecal volatile organic compounds, fecal volatile organic compounds under chemotherapy and final fecal volatile organic compounds) and breath organic volatile compounds (initial breath organic compounds, breath volatile organic compounds under chemotherapy and final breath volatile organic compounds).
  Samples will be taken after verifying diagnosis before initiation of chemotherapy, 1 week after completion of each cycle and 3 weeks after the end of chemotherapy.
  Interventions: Diagnostic Test: Initial fecal microbiome; Diagnostic Test: Initial fecal volatile organic compounds; Diagnostic Test: Initial breath volatile organic compounds; Diagnostic Test: Microbiome under chemotherapy; Diagnostic Test: Fecal volatile organic compounds under chemotherapy; Diagnostic Test: Breath volatile organic compounds under chemotherapy; Diagnostic Test: Final microbiome; Diagnostic Test: Final fecal volatile organic compounds; Diagnostic Test: Final breath volatile organic compounds
- Control group (Other): 10 children without gastro-intestinal or pulmonary disease as age and sex matched controls to the neuroblastoma group. Patients will be recruited from paediatric surgery. Inclusion after informed consent.
  Sampling of fecal microbiome (initial fecal microbiome), fecal volatile organic compounds (initial fecal volatile organic compounds) and breath organic volatile compounds (initial breath volatile organic compounds).
  Samples will be taken as age and sex matched controls for the neuroblastoma group. Sampling will be done once after obtaining informed consent.
  Interventions: Diagnostic Test: Initial fecal microbiome; Diagnostic Test: Initial fecal volatile organic compounds; Diagnostic Test: Initial breath volatile organic compounds

INTERVENTIONS:
Diagnostic Test: Initial fecal microbiome — Stool sampling for fecal microbiome analysis by 16S rDNA pyrosequencing. Neuroblastoma group and Control group.
Diagnostic Test: Initial fecal volatile organic compounds — Volatile organic compound analysis of stool samples by gas chromatography/mass spectroscopy Neuroblastoma group and Control group.
Diagnostic Test: Initial breath volatile organic compounds — Breath sampling for organic compound analysis by gas chromatography/mass spectroscopy Neuroblastoma group and Control group.
Diagnostic Test: Microbiome under chemotherapy — Stool sampling under chemotherapy of children in neuroblastoma group (1 sample 1 week after completion of each chemotherapy cycle). Chemotherapy according to Société Internationale d´Onclogie Pediatrique Neuroblastoma Group (SIOPEN) guidelines
  Arms: Neuroblastoma group
Diagnostic Test: Fecal volatile organic compounds under chemotherapy — Stool sampling under chemotherapy of children in neuroblastoma group (1 sample 1 week after completion of each chemotherapy cycle). Chemotherapy according to SIOPEN guidelines.
  Neuroblastoma group
  Arms: Neuroblastoma group
Diagnostic Test: Breath volatile organic compounds under chemotherapy — Breath sampling under chemotherapy of children in neuroblastoma group (1 sample 1 week after completion of each chemotherapy cycle). Chemotherapy according to SIOPEN guidelines.
  Neuroblastoma group
  Arms: Neuroblastoma group
Diagnostic Test: Final microbiome — Stool sampling 3 weeks after completion of chemotherapy Neuroblastoma group
  Arms: Neuroblastoma group
Diagnostic Test: Final fecal volatile organic compounds — Stool sampling 3 weeks after completion of chemotherapy Neuroblastoma group
  Arms: Neuroblastoma group
Diagnostic Test: Final breath volatile organic compounds — Breath sampling 3 weeks after completion of chemotherapy Neuroblastoma group
  Arms: Neuroblastoma group

SUMMARY:
Background: Malignant tumors may lead to a catabolic state with loss of muscle and adipose tissue. The full picture of catabolism is termed cachexia and is associated with significant morbidity and mortality of cancer patients. Although the full picture is rarely observed up to 50% of children with cancer suffer from significant malnourishment. Additionally to tumor-induced catabolism, side-effects of chemotherapy may be problematic for the patients. In this regard up to 60% of children suffer from gastrointestinal mucositis presenting with nausea, vomiting, diarrhea or constipation and abdominal pain. In the worst case, mucositis may lead to bacterial translocation with life-threatening inflammatory response. Clinically this may require a reduction of the dosage or the number of chemotherapy cycles resulting in reduced effectivity. Up to now the therapy of mucositis is only symptomatic. Recent research of the applicant has shown a significant reduction of Lactobacilli in mice with neuroblastoma (a malignant childhood tumor). The dysbiosis was associated with catabolism, increased gut permeability and inflammation. Astonishingly, chemotherapy alone also leads to a significant reduction of Lactobacilli compared to sham mice, which may be linked to the development of mucositis clinically. Overall, the intestinal microbiome seems to play an essential role in the development of tumor-associated catabolism and chemotherapy-induced mucositis.

Aim: The aim of this project is to determine if the changes in the intestinal microbiome observed in mice can also be seen in children with neuroblastoma.

Methods: One part of the study will include 10 children with neuroblastoma (inclusion after verification of the diagnosis) and 10 healthy controls. The fecal microbiome will be determined by 16S-ribosomal deoxyribonucleic acid (rDNA) pyrosequencing. Volatile organic compounds in the breath will be sampled and measured by Gas Chromatography/Mass Spectroscopy. A basic science human work package will address the question if there are differences.

In the second part serial investigations in children with neuroblastoma will assess whether or not these patients show alterations of the intestinal microbiome under chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-8 years
* Neuroblastoma group: verified neuroblastoma
* Control group: absence of pulmonary or gastro-intestinal disease
* Written parental informed consent obtained

Exclusion Criteria:

* Active gastro-intestinal or pulmonary disease
* Antibiotic or probiotic treatment within 3 weeks before sampling
* Negative parental informed consent

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of alpha and beta diversity, relative abundance of fecal bacteria at different levels (phylum, class, order, family and genus levels) between neuroblastoma and control group | Neuroblastoma group: within 48h after diagnosis, before initiation of chemotherapy. Control group: within 24h after obtaining informed consent.
  Alpha and beta diversity, relative bacterial abundance at different levels in percent.
Change of alpha and beta diversity, relative abundance of fecal bacteria at different levels (phylum, class, order, family and genus levels) under chemotherapy in the neuroblastoma group | Within 48h after diagnosis, before initiation of chemotherapy; 1 week after each chemotherapy cycle and 3 weeks after the end of chemotherapy.
  Alpha and beta diversity, relative bacterial abundance at different levels in percent.

SECONDARY OUTCOMES:
Difference of anthropometric data between neuroblastoma and control group. | Neuroblastoma group: within 48h after diagnosis. Control group: within 24h after obtaining informed consent.
  Body weight (in kg) and height (in m) will be determined to calculate the body mass index (BMI in kg/m^2).
Change of anthropometric data under chemotherapy in the neuroblastoma group | Within 48h after diagnosis, before initiation of chemotherapy; 7 days after completion of each chemotherapy cycle and 3 weeks after the end of chemotherapy.
  Body weight (in kg) and height (in m) will be determined to calculate the Body mass index (BMI in kg/m^2).
Change of mucositis score under chemotherapy in the neuroblastoma group. | Within 48h after diagnosis, before initiation of chemotherapy; 7 days after completion of each chemotherapy cycle and 3 weeks after the end of chemotherapy.
  Assessment of the mucositis score according to the WHO criteria (WHO handbook for reporting results of cancer Treatment; WHO Offset publication no 48) The score contains 5 subitems which are evaluated separately. At the end a total score is derived by adding the results of all items.
  Subitem 1: oral mucosa; range 0 (best) to 4 (worst) Subitem 2: nausea and vomiting; range from 0 (best) to 4 (worst) Subitem 3: diarrhea; range from 0 (best) to 4 (worst) Subitem 4: constipation; range from 0 (best) to 4 (worst) Subitem 5: abdominal pain; range from 0 (best) to 4 (worst)
Difference of breath volatile organic compounds between neuroblastoma and control group. | Neuroblastoma group: within 48h after diagnosis. Control group: within 24h after obtaining informed consent.
  Volatile organic compounds in ppb in the exhaled breath.
Difference of stool volatile organic compounds between neuroblastoma and control group. | Neuroblastoma group: within 48h after diagnosis. Control group: within 24h after obtaining informed consent.
  Volatile organic compounds in ppb in stool samples.
Change of breath volatile organic compounds under chemotherapy in the neuroblastoma group. | Within 48h after diagnosis, before initiation of chemotherapy; 1 week after each chemotherapy cycle and 3 weeks after the end of chemotherapy.
  Volatile organic compounds in ppb in the exhaled breath.
Change of stool volatile organic compounds under chemotherapy in the neuroblastoma group. | Within 48h after diagnosis, before initiation of chemotherapy; 1 week after each chemotherapy cycle and 3 weeks after the end of chemotherapy.
  Volatile organic compounds in ppb in stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Castellani, MD, Principal Investigator — Department of Paediatric and Adolescent Surgery, Medical University of Graz, Austria
Locations (1):
- Department of Paediatric and Adolescent Surgery, Medical University of Graz, Austria, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No